CLINICAL TRIAL: NCT03395080
Title: A Phase 2 Study Evaluating the Efficacy and Safety of DKN-01 as a Monotherapy or in Combination With Paclitaxel in Patients With Recurrent Epithelial Endometrial, Epithelial Ovarian Cancer, or Carcinosarcoma
Brief Title: A Study of DKN-01 as a Monotherapy or in Combination With Paclitaxel in Patients With Recurrent Epithelial Endometrial or Epithelial Ovarian Cancer or Carcinosarcoma
Acronym: P204
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leap Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEK-DKK1-P204
Record Dates: First submitted 2018-01-02; First posted 2018-01-10 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2023-05

CONDITIONS: Endometrial Cancer; Uterine Cancer; Ovarian Cancer; Carcinosarcoma
Keywords: epithelial histology; Wnt pathway; DKK1; endometrial; uterine; ovarian; carcinosarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Ovarian Neoplasms; Carcinosarcoma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- DKN-01 monotherapy in recurrent EEC (Experimental): 300mg DKN-01 monotherapy in recurrent EEC
  Interventions: Drug: 300mg DKN-01
- DKN-01+paclitaxel in recurrent EEC (Experimental): 300mg DKN-01+paclitaxel in recurrent EEC
  Interventions: Drug: Paclitaxel; Drug: 300mg DKN-01
- DKN-01 monotherapy in recurrent EOC (Experimental): 300mg DKN-01 monotherapy in recurrent EOC
  Interventions: Drug: 300mg DKN-01
- DKN-01+paclitaxel in recurrent EOC (Experimental): 300mg DKN-01+paclitaxel in recurrent EOC
  Interventions: Drug: Paclitaxel; Drug: 300mg DKN-01
- DKN-01 monotherapy in carcinosarcoma (Experimental): 600mg DKN-01 monotherapy in carcinosarcoma
  Interventions: Drug: 600mg DKN-01
- DKN-01 +paclitaxel in carcinosarcoma (Experimental): 600mg DKN-01 +paclitaxel in carcinosarcoma
  Interventions: Drug: Paclitaxel; Drug: 600mg DKN-01

INTERVENTIONS:
Drug: Paclitaxel — Administered by IV infusion
  Other Names: Taxol
  Arms: DKN-01 +paclitaxel in carcinosarcoma; DKN-01+paclitaxel in recurrent EEC; DKN-01+paclitaxel in recurrent EOC
Drug: 300mg DKN-01 — Administered by IV infusion
  Arms: DKN-01 monotherapy in recurrent EEC; DKN-01 monotherapy in recurrent EOC; DKN-01+paclitaxel in recurrent EEC; DKN-01+paclitaxel in recurrent EOC
Drug: 600mg DKN-01 — Administered by IV infusion
  Arms: DKN-01 +paclitaxel in carcinosarcoma; DKN-01 monotherapy in carcinosarcoma

SUMMARY:
A Phase 2 Study Evaluating the Efficacy and Safety of DKN-01 as a Monotherapy or in Combination with Paclitaxel in Patients With Recurrent Epithelial Endometrial Cancer, Epithelial Ovarian Cancer, or Carcinosarcoma

DETAILED DESCRIPTION:
This study employs a "basket" design to concurrently investigate DKN-01 as monotherapy and in combination with paclitaxel in patients with recurrent epithelial endometrial cancer (EEC), epithelial ovarian cancer (EOC), or carcinosarcoma (malignant mixed Mullerian tumor [MMMT]. Thus, 6 distinct patient groups are being independently investigated:

1. 300mg DKN-01 monotherapy in recurrent EEC (Group 1)
2. 300mg DKN-01+paclitaxel in recurrent EEC (Group 2)
3. 300mg DKN-01 monotherapy in recurrent EOC (Group 3)
4. 300mg DKN-01+paclitaxel in recurrent EOC (Group 4)
5. 600mg DKN-01 monotherapy in recurrent carcinosarcoma (MMMT) (Group 5)
6. 600mg DKN-01+paclitaxel in recurrent carcinosarcoma (MMMT) (Group 6)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis:

   1. Epithelial Endometrial Cancer: histologically confirmed diagnosis (by either primary surgical specimen or biopsy for recurrence) of recurrent previously treated EEC.
   2. Epithelial Ovarian Cancer: histologically confirmed diagnosis (by either primary surgical specimen or biopsy for recurrence) of recurrent platinum-resistant/refractory EOC, primary peritoneal, or fallopian tube cancer (i.e., disease recurrence within 6 months of completion of or progression during platinum-based chemotherapy).
   3. Carcinosarcoma/Malignant Mixed Mullerian Tumors: histologically confirmed diagnosis (by either primary surgical specimen or biopsy for recurrence) of recurrent uterine or ovarian carcinosarcoma (MMMT). Patients must have had only 1 prior chemotherapeutic regimen for management of carcinosarcoma that may have been included chemotherapy (including in adjuvant setting), chemotherapy and radiotherapy, and/or consolidation/maintenance therapy.
2. Refractory or intolerant to at least one prior standard therapy(ies) for metastatic or locally advanced disease (see Inclusion Criterion #1c for Groups 5-6).

   1. If prior therapy consisted of palliative chemoradiation therapy, it will be considered one line of therapy.
   2. Prior treatment with paclitaxel as part of definitive therapy regimen is acceptable, provided the patient is not intolerant of paclitaxel.
   3. Patients who are not eligible to receive paclitaxel will be allowed to receive single agent DKN-01.
3. Tumor tissue for mandatory pre-treatment and on-treatment biopsies.
4. One or more tumors measurable on radiographic imaging as defined by RECIST 1.1.
5. Ambulatory and ≥18 years of age.
6. ECOG performance status (PS) of 0 or 1

   a. ECOG PS of 2 may be eligible upon the review and approval of the Medical Monitor.
7. Estimated life expectancy of at least 3 months, in the judgment of the Investigator.
8. Disease-free of active second/secondary or prior malignancies for ≥2 years with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix or breast.
9. Acceptable liver, renal, hematologic and coagulation function
10. Females of child bearing potential and male partners of female patients must agree to use adequate contraception during the study and for 6 months after their last dose of study drug.
11. Reliable and willing to make themselves available for the duration of the study and are willing to follow study-specific procedures.
12. Provided written informed consent prior to any study-specific procedures.

Exclusion Criteria:

1. Patients with the following pure histologies of endometrial or ovarian cancer are not eligible for enrollment: germ cell, sex cord stroma, or sarcoma.
2. New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
3. Fridericia-corrected QT interval (QTcF) > 470 msec (female) or history of congenital long QT syndrome.
4. Active, uncontrolled bacterial, viral, or fungal infections, within 7 days of study entry requiring systemic therapy.
5. Known to be human immunodeficiency virus (HIV) positive, have hepatitis B surface antigen (HBSAg), or hepatitis C antibodies (HCAb), unless hepatitis C virus ribonucleic acid (HCV RNA) undetected/negative.
6. History of major organ transplant (i.e., heart, lungs, liver, or kidney).
7. History of autologous/allogenic bone marrow transplant.
8. Serious nonmalignant disease
9. Pregnant or nursing.
10. History of osteonecrosis of the hip or have evidence of structural bone abnormalities in the proximal femur on MRI scan that are symptomatic and clinically significant.
11. Symptomatic central nervous system (CNS) malignancy or metastasis.
12. Known osteoblastic bony metastasis
13. Treatment with surgery or chemotherapy within 21 days prior to study entry (42 days for nitrosoureas or mitomycin C)
14. Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to study entry.
15. Clinically significant peripheral neuropathy at the time of study entry. Patients with pre-existing peripheral neuropathy will be allowed to receive single agent DKN-01
16. History of hypersensitivity reactions to paclitaxel or other drugs formulated in Cremophor® EL (polyoxyethylated castor oil). Patients who exhibit these hypersensitivities will be eligible to receive single agent DKN-01
17. Prior radiation therapy within 14 days prior to study entry
18. Currently receiving any other investigational agent or received an investigational agent within last 30 days of study entry.
19. Previously treated with an anti-DKK1 therapy
20. Significant allergy to a pharmaceutical therapy that, in the opinion of the Investigator, poses an increased risk to the patient
21. Active substance abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gender identity
Enrollment: 111 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Sirard, Study Director — Leap Therapeutics
Locations (17):
- United States (17):
  - University of Alabama, Birmingham, Alabama
  - HonorHealth, Scottsdale, Arizona
  - Florida Cancer Specialists & Research Institute, West Palm Beach, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - HCA Midwest Health System Clinical Research, Kansas City, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Hilliard, Ohio
  - Stephenson Cancer Center - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The University of Tennessee West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Arend R, Dholakia J, Castro C, Matulonis U, Hamilton E, Jackson CG, LyBarger K, Goodman HM, Duska LR, Mahdi H, ElNaggar AC, Kagey MH, Liu A, Piper D, Barroilhet LM, Bradley W, Sachdev J, Sirard CA, O'Malley DM, Birrer M. DKK1 is a predictive biomarker for response to DKN-01: Results of a phase 2 basket study in women with recurrent endometrial carcinoma. Gynecol Oncol. 2023 May;172:82-91. doi: 10.1016/j.ygyno.2023.03.013. Epub 2023 Mar 29. PMID 37001446

RESULTS

PARTICIPANT FLOW:
Groups:
- DKN-01 Monotherapy in Recurrent EEC: 300mg DKN-01 monotherapy in recurrent EEC. DKN-01 administered by IV infusion.
- DKN-01+Paclitaxel in Recurrent EEC: 300mg DKN-01+paclitaxel in recurrent EEC. DKN-01 administered by IV infusion.
- DKN-01 Monotherapy in Recurrent EOC: 300mg DKN-01 monotherapy in recurrent EOC. DKN-01 administered by IV infusion.
- DKN-01+Paclitaxel in Recurrent EOC: 300mg DKN-01+paclitaxel in recurrent EOC. DKN-01and paclitaxel administered by IV infusion.
- DKN-01 300mg Monotherapy in Carcinosarcoma: 300mg DKN-01 monotherapy in carcinosarcoma. DKN-01 administered by IV infusion.
- DKN-01 600mg Monotherapy in Carcinosarcoma: 600mg DKN-01 monotherapy in carcinosarcoma. DKN-01 administered by IV infusion.
- DKN-01 300mg + Paclitaxel in Carcinosarcoma: 300mg DKN-01 + paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 600 mg + Paclitaxel in Carcinosarcoma: 600mg DKN-01 + paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
Period: Overall Study
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01+Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01+Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600 mg + Paclitaxel in Carcinosarcoma
Started (Number Started is the Safety Analysis Set defined as all subjects who received >= 1 administration of assigned study treatment (DKN-01 or paclitaxel).Subjects with carcinosarcoma were initially enrolled in the EEC group to receive monotherapy or DKN-01+paclitaxel, but as part of a subsequent protocol amendment, carcinosarcoma subjects were enrolled & received 600mg DKN-01 or 600mg DKN-01+paclitaxel. Results are reported by disease type and treatment received.) | 29 | 24 | 14 | 19 | 1 | 8 | 4 | 12
Completed (Number Completed is the Evaluable Analysis Set defined as all subjects who received any amount of DKN-01 and had at least 1 evaluated post-baseline RECIST assessment or were discontinued due to death.) | 26 | 21 | 13 | 19 | 1 | 8 | 4 | 10
Not Completed | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- DKN-01+Paclitaxel in Recurrent EEC: 300mg DKN-01+paclitaxel in recurrent EEC. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01+Paclitaxel in Recurrent EOC: 300mg DKN-01+paclitaxel in recurrent EOC. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 300mg+Paclitaxel in Carcinosarcoma: 300mg DKN-01 +paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 600mg+Paclitaxel in Carcinosarcoma: 600mg DKN-01 +paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
- Total: Total of all reporting groups
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01+Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01+Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg+Paclitaxel in Carcinosarcoma | DKN-01 600mg+Paclitaxel in Carcinosarcoma | Total
Number analyzed (Participants) | 29 | 24 | 14 | 19 | 1 | 8 | 4 | 12 | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 12 | 5 | 10 | 1 | 2 | 2 | 8 | 59
  >=65 years | 10 | 12 | 9 | 9 | 0 | 6 | 2 | 4 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 14 | 19 | 1 | 8 | 4 | 12 | 111
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 7
  Not Hispanic or Latino | 25 | 23 | 14 | 18 | 1 | 7 | 4 | 10 | 102
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 2 | 3 | 0 | 1 | 0 | 0 | 8
  White | 27 | 21 | 12 | 16 | 1 | 7 | 4 | 9 | 97
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Objective Response Rate (ORR) in EEC or EOC Patients
Description: Best overall response of Complete Response (CR; disappearance of all target lesions, any pathological lymph nodes whether target or non-target must have reduction in short axis to <10mm) or Partial Response (PR; at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1)
Time Frame: Baseline to study completion (approximately 6 months)
Population: Evaluable Analysis Set (EAS), all subjects who received any amount of DKN-01 and had at least 1 evaluated post-baseline RECIST assessment or were discontinued due to death.
Measure: Number; unit: participants
Groups:
- DKN-01 + Paclitaxel in Recurrent EEC: 300mg DKN-01+paclitaxel in recurrent EEC. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 + Paclitaxel in Recurrent EOC: 300mg DKN-01+paclitaxel in recurrent EOC. DKN-01 and paclitaxel administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC
Number analyzed (Participants) | 26 | 21 | 13 | 19
participants
  ORR | 2 | 0 | 0 | 0
  Complete Response | 1 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 0
  Stable Disease | 9 | 12 | 6 | 13
  Progressive Disease | 15 | 9 | 7 | 6

2. Primary Outcome: Number of Subjects With Objective Response Rate (ORR) in Carcinosarcoma (MMMT) Patients
Description: as for outcome 1
Time Frame: Baseline to study completion (approximately 6 months)
Population: Evaluable Analysis Set, all subjects who received any amount of DKN-01 and had at least 1 evaluated post-baseline RECIST assessment or were discontinued due to death.
Measure: Number; unit: participants
Groups:
- DKN-01 600mg + Paclitaxel in Carcinosarcoma: 600mg DKN-01 + paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
Arm/Group | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 1 | 8 | 4 | 10
participants
  Confirmed ORR | 0 | 0 | 1 | 1
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 1 | 1
  Stable Disease | 1 | 1 | 0 | 4
  Progressive Disease | 0 | 7 | 3 | 5

3. Secondary Outcome: Number of Subjects With Objective Disease Control Rate (ODCR) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Objective Disease Control Rate (ODCR) was defined as the percentage of subjects with a Best Overall Response of Complete Response (CR; disappearance of all target lesions, any pathological lymph nodes whether target or non-target must have reduction in short axis to <10mm), Partial Response (PR; at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters), or Stable Disease (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify as Progressive Disease) as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1)
Time Frame: Baseline to study completion (approximately 6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 26 | 21 | 13 | 19 | 1 | 8 | 4 | 10
Participants | 11 | 12 | 6 | 13 | 1 | 1 | 1 | 5

4. Secondary Outcome: Overall Survival (OS) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Overall Survival (OS) is defined as the time from first dose of study drug until date of death due to any cause.
Time Frame: Baseline to study completion (maximum 17.6 months)
Population: Full Analysis Set (FAS), all subjects who received any amount of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 29 | 24 | 14 | 19 | 1 | 8 | 4 | 12
months | 12.2 [4.6 to NA] — NA=Not Estimable. Data are not estimable due to insufficient number of participants with events. | 10.1 [6.5 to 13.6] | 10.8 [5.7 to 17.6] | 11.9 [6.6 to NA] — NA=Not Estimable. Data are not estimable due to insufficient number of participants with events. | NA [NA to NA] — Data are not estimable due to insufficient number of participants with events. | 8.4 [1.3 to NA] — NA=Not Estimable. Data are not estimable due to insufficient number of participants with events. | 7.3 [5.3 to NA] — NA=Not Estimable. Data are not estimable due to insufficient number of participants with events. | 5.7 [1.6 to NA] — NA=Not Estimable. Data are not estimable due to insufficient number of participants with events.

5. Secondary Outcome: Progression-free Survival (PFS) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Progression-free survival (PFS) is defined as time from first dose of study drug to first documentation of PD (per RECIST 1.1) or death due to any cause.
Time Frame: Baseline to study completion (maximum 7.1 months)
Population: Full Analysis Set (FAS), all subjects who received any amount of DKN-01.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DKN-01 600mg Monotherapy in Carcinosarcoma: 600mg DKN-01 onotherapy in carcinosarcoma. DKN-01 administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 29 | 24 | 14 | 19 | 1 | 8 | 4 | 10
months | 1.8 [1.7 to 5.5] | 3.8 [1.8 to 5.4] | 2.1 [1.6 to 3.5] | 3.6 [1.8 to 7.1] | 11.6 [NA to NA] — NA=not estimable. Data are not estimable due to insufficient number of participants with events. | 1.6 [0.5 to 7.9] | 2.0 [1.8 to 5.5] | 1.9 [0.9 to 4.0]

6. Secondary Outcome: Duration of Response (DoR) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Duration of Response (DoR) includes only patients that have responded with an objective disease response (PR or CR) and is defined as the time from the first tumor assessment that supports the patient's objective disease response to the time of PD or death due to any cause.
Time Frame: Baseline to study completion (approximately 11 months)
Population: Number of participants analyzed only includes the responders in each group.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DKN-01 + Paclitaxel in Eecurrent EOC: 300mg DKN-01+paclitaxel in recurrent EOC. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 300mg Monotherapy in Carcinosarcoma: 300mg DKN-01 in carcinosarcoma. DKN-01 administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Eecurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1
months | NA [NA to NA] — NA = Insufficient number of participants with events. 2 subjects with responses, but only one with an event, Median duration of response could not be estimated as 1 of the 2 subjects response had not had a progression event, therefore the 95% CIs are not estimable. 1 patient remains in response at end of study. |  |  |  |  |  | 3.7 [NA to NA] — PR was reported for 1 subject with a progression event therefore no CIs are estimable | NA [NA to NA] — Insufficient number of participants with events. Median duration of response could not be estimated as the 1 subject with PR had not had a progression event.

7. Secondary Outcome: Duration of Complete Response (DoCR) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Number of participants analyzed only includes patients with a CR and is otherwise defined and analyzed similar to DoR.
Time Frame: Baseline to study completion (approximately 11 months)
Population: Number of participants analyzed only includes patients who have responded with an objective disease response (CR).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DKN-01 + Paclitaxel in Recurrent EEC: 300mg DKN-01 + paclitaxel in recurrent EEC. DKN-01 and paclitaxel administered by IV infusion.
- DKN-01 + Paclitaxel in Recurrent EOC: 300mg DKN-01 + paclitaxel in recurrent EOC. DKN-01 and paclitaxel administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinosarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
months | NA [NA to NA] — Insufficient number of participants with events. |  |  |  |  |  |  |

8. Secondary Outcome: Duration of Clinical Benefit (DoCB) in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Description: Duration of Clinical Benefit (DoCB) includes patients with a Best Overall Response of CR, PR, or SD and is defined as the time from the first tumor assessment of CR, PR or SD to the time of PD or death due to any cause.
Time Frame: Baseline to study completion (approximately 13.1 months)
Population: Number of participants analyzed only includes patients who had CR, PR, or SD.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- DKN-01 300mg + Paclitaxel in Carcinsarcoma: 300mg DKN-01 + paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01 + Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01 + Paclitaxel in Recurrent EOC | DKN-01 300mg Monotherapy in Carcinosarcoma | DKN-01 600mg Monotherapy in Carcinosarcoma | DKN-01 300mg + Paclitaxel in Carcinsarcoma | DKN-01 600mg + Paclitaxel in Carcinosarcoma
Number analyzed (Participants) | 11 | 12 | 6 | 13 | 1 | 1 | 1 | 5
months | 4.7 [1.2 to 9.2] | 3.8 [2.0 to 4.2] | 1.9 [1.7 to 13.1] | 3.9 [1.8 to 5.6] | NA [NA to NA] — Subject had a progression event; the Kaplan-Meier estimated median duration of clinical benefit times was not estimable. | 6.0 [NA to NA] — NA = not estimable. Data are not estimable due to insufficient number of participants with events. | 3.7 [NA to NA] — NA = not estimable. Data are not estimable due to insufficient number of participants with events. | 2.2 [1.9 to NA] — NE = not estimable. Data are not estimable due to insufficient number of participants with events.

9. Other Pre Specified Outcome: Number of Subjects With Response to Therapy in Patients With and Without Activating β-catenin Mutations and/or Wnt Signaling Genetic Alterations in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Dickkopf-1 (DKK1) Concentration in Serum and Plasma Relative to Safety and Efficacy Outcomes in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT).
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Subjects With Adverse Drug Reactions and Toxicities as Evaluated by NCI CTCAE v5.0 of DKN-01 600 mg +/- Paclitaxel in Patients With Recurrent Carcinosarcoma (MMMT) in Carcinosarcoma (MMMT) Patients
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Maximum Plasma Concentration (Cmax)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Time Taken to Reach the Maximum Plasma Concentration (Tmax)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Area Under the Curve (AUC)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Number of Subjects With Adverse Drug Reactions and Toxicities as Evaluated by NCI CTCAE v4.03 as DKN-01 as Monotherapy or in Combination With Paclitaxel in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Number of Subjects With Adverse Drug Reactions and Toxicities to Study Treatment Regimen in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT) as Evaluated by NCI CTCAE v5.0
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Concentration of DKN-01 Antibodies in Human Serum in Patients With Recurrent EEC or EOC or Carcinosarcoma (MMMT)
Time Frame: Baseline to study completion (approximately 6 months)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The Safety Analysis Set is all subjects who received greater than or equal to 1 administration of assigned study treatment (DKN-01 or paclitaxel). Subjects were followed for treatment emergent adverse events (AE), defined as any AE with an onset or worsening of a pre-existing condition on or after the first dose of the study drug through 30 days following the last dose of study drug, up to approximately 2 years.
Description: Adverse events and serious adverse events reported are those that started or worsened after the first dose of study treatment and within 30 days after the last study treatment dose.
Groups:
- 300mg DKN-01 Monotherapy in Carcinosarcoma: 300mg DKN-01 monotherapy in carcinosarcoma. DKN-01 administered by IV infusion.
- 600mg DKN-01 Monotherapy in Carcinosarcoma: 600mg DKN-01 monotherapy in carcinosarcoma. DKN-01 administered by IV infusion.
- 300mg DKN-01+Paclitaxel in Carcinosarcoma: 300mg DKN-01+paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
- 600mg DKN-01+Paclitaxel in Carcinosarcoma: 600mg DKN-01+paclitaxel in carcinosarcoma. DKN-01 and paclitaxel administered by IV infusion.
Arm/Group | DKN-01 Monotherapy in Recurrent EEC | DKN-01+Paclitaxel in Recurrent EEC | DKN-01 Monotherapy in Recurrent EOC | DKN-01+Paclitaxel in Recurrent EOC | 300mg DKN-01 Monotherapy in Carcinosarcoma | 600mg DKN-01 Monotherapy in Carcinosarcoma | 300mg DKN-01+Paclitaxel in Carcinosarcoma | 600mg DKN-01+Paclitaxel in Carcinosarcoma
All-Cause Mortality (participants affected / at risk) | 14/29 | 16/24 | 11/14 | 12/19 | 0/1 | 4/8 | 2/4 | 8/12
Serious Adverse Events (participants affected / at risk) | 8/29 | 13/24 | 1/14 | 6/19 | 1/1 | 2/8 | 0/4 | 6/12
Other Adverse Events (participants affected / at risk) | 29/29 | 24/24 | 13/14 | 19/19 | 1/1 | 8/8 | 4/4 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DKN-01 Monotherapy in Recurrent EEC (N=29) | DKN-01+Paclitaxel in Recurrent EEC (N=24) | DKN-01 Monotherapy in Recurrent EOC (N=14) | DKN-01+Paclitaxel in Recurrent EOC (N=19) | 300mg DKN-01 Monotherapy in Carcinosarcoma (N=1) | 600mg DKN-01 Monotherapy in Carcinosarcoma (N=8) | 300mg DKN-01+Paclitaxel in Carcinosarcoma (N=4) | 600mg DKN-01+Paclitaxel in Carcinosarcoma (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | DKN-01 Monotherapy in Recurrent EEC (N=29) | DKN-01+Paclitaxel in Recurrent EEC (N=24) | DKN-01 Monotherapy in Recurrent EOC (N=14) | DKN-01+Paclitaxel in Recurrent EOC (N=19) | 300mg DKN-01 Monotherapy in Carcinosarcoma (N=1) | 600mg DKN-01 Monotherapy in Carcinosarcoma (N=8) | 300mg DKN-01+Paclitaxel in Carcinosarcoma (N=4) | 600mg DKN-01+Paclitaxel in Carcinosarcoma (N=12)
Anaemia (Blood and lymphatic system disorders) | 7 | 13 | 2 | 3 | 0 | 0 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 5 | 1 | 5 | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 10 | 8 | 8 | 0 | 1 | 2 | 4
Constipation (Gastrointestinal disorders) | 5 | 6 | 4 | 2 | 0 | 1 | 0 | 3
Vomiting (Gastrointestinal disorders) | 7 | 6 | 2 | 5 | 0 | 1 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 3 | 6 | 0 | 2 | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 4 | 6 | 3 | 2 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 7 | 3 | 10 | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal wall cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 4 | 0 | 1 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 13 | 11 | 9 | 7 | 0 | 2 | 0 | 7
Oedema peripheral (General disorders) | 4 | 8 | 0 | 4 | 0 | 1 | 0 | 2
Chills (General disorders) | 2 | 3 | 0 | 2 | 1 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 3 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medical device site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1 | 0 | 0/0 | 0/0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 | 6 | 0 | 6 | 0 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 2
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection eterococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 2 | 0 | 0 | 1 | 0 | 1
Blood cholesterol increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 3 | 0 | 1 | 0 | 1 | 0 | 0
Activate partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 2 | 2 | 0 | 1 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 3 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 4 | 1 | 3 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6 | 1 | 2 | 0 | 0 | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2 | 3 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 2 | 0 | 1 | 2 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 1 | 0 | 0 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0/0 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0/0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 4 | 3 | 4 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 5 | 5 | 0 | 1 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 6 | 1 | 0 | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 4 | 1 | 3 | 0 | 1 | 0 | 3
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Parosmia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 0 | 3 | 0 | 1 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restless leg syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 3
Confusional state (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 3 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 2 | 0 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 8 | 0 | 8 | 1 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Dermatitus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 1 | 1 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03395080/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT03395080/SAP_001.pdf